CLINICAL TRIAL: NCT01270893
Title: A Two-Arm Study of Preoperative Nilotinib for Patients With Resectable or Potentially Resectable Gastrointestinal Stromal Tumor (GIST)
Brief Title: Tasigna Neoadjuvant Gastrointestinal Stromal Tumor (GIST)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No particapnt recruitment.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0722
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal stromal tumor; GIST; Nilotinib; AMN107; Tasigna
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nilotinib and Surgical Resection (Experimental)
  Interventions: Drug: Nilotinib
- Nilotinib and Potential Resection (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 400 mg by mouth twice a day for 7 days. Patients on Arm 2 will continue to receive Nilotinib until they have disease progression or are resectable.
  Other Names: AMN107; Tasigna

SUMMARY:
The goal of this clinical research study is to learn if Tasigna® (nilotinib) can cause tumor cells to shrink and/or die in patients with GIST who are scheduled for surgery or may be eligible for surgery. The safety of this drug will be studied. Researchers also want to use imaging scans to study the changes in tumor size that may be caused by using nilotinib.

DETAILED DESCRIPTION:
GIST is a rare cancer known as a soft-tissue sarcoma that forms in the gastrointestinal (GI) tract and may spread to other parts of the body. However, sometimes GIST stays in the GI tract where it may possibly be removed by surgery. While some chemotherapy drugs, such as imatinib mesylate, are effective in shrinking or controlling GIST, some types of GIST tumors do not respond to imatinib. Researchers want to find out if nilotinib (a drug similar to imatinib) causes GIST cells to die, so that the tumors shrink enough to be removed by surgery.

The Study Drugs:

Nilotinib is designed to prevent cells from multiplying by causing tumor cells to shrink and/or die. This may prevent the cancer from growing.

Study Arms and Study Drug Administration:

If you are found to be eligible to take part in this study, a surgeon from M. D. Anderson will check your imaging scans to decide if the tumor can be surgically removed.

Participants in this research study will be assigned to either Arm 1 or Arm 2, based on whether the tumor is able to be removed by surgery at this point.

Arm 1:

If the surgeon thinks the tumor is able to be removed during surgery, you will be assigned to Arm 1. You will receive nilotinib pills by mouth 2 times a day for 7 days. You will receive a pill diary and will be shown how to record the date and time for each dose received.

After the week of nilotinib therapy, you will be scheduled to have the GIST removed during surgery. Tumor tissue that is removed during surgery will be used for research testing. Some of these tests will help researchers learn how effectively nilotinib kills tumor cells. Your DNA and RNA (the genetic material in your cells) will also be collected from these tissue samples and used to help researchers understand how these tumor cells survive, divide, and die as a result of nilotinib.

After 4-6 weeks of recovery time after surgery, you will receive standard of care treatment off-study.

An assigned research nurse will see you at each clinic visit and will serve as the first contact for any questions or concerns. During the course of this study, you will be asked to report any serious problems or concerns at each study visit. If you have concerns or questions between each study visits, you may contact your study nurse through the Sarcoma Center at M. D. Anderson.

Arm 1 Study Visits:

Participants in Arm 1 will have the following tests and procedures performed:

On Day -7, you will begin taking nilotinib.

On Day -1:

* You will have a dynamic CT scan within 36 hours before surgery to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 0, you will have surgery to remove the GIST.

On Day 56:

* You will be asked about your health, any drugs you may be taking, and any side effects you may have experienced.
* You will have a physical exam, including measurement of vital signs and weight.
* Your performance status will be recorded.
* You will have a chest x-ray.
* You will have a standard CT scan or an MRI scan to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

Every 3 months:

* You will be asked about your health, any drugs you may be taking, and any side effects you may have experienced.
* You will have a physical exam, including measurement of vital signs and weight.
* Your performance status will be recorded.
* You will have a standard CT scan or an MRI scan to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

Arm 2:

If the surgeon thinks the tumor is not able to be surgically removed at this time, or that the tumor needs to shrink before it can be removed during surgery, you will be assigned to Arm 2. You will receive nilotinib pills by mouth 2 times a day for 7 days. You will receive a pill diary and will be shown how to record the date and time for each dose received.

After the week of nilotinib therapy, you will be scheduled to have a biopsy on what is counted as Day 0 on your pill diary. After 7 days of recovery from the biopsy, you will continue receiving nilotinib on the same schedule (2 times a day by mouth).

After 8 weeks of nilotinib therapy, you will have more scans performed to measure the size of the tumor. These scans will include a CT scan of your abdomen or pelvis. You may have a magnetic resonance imaging (MRI) scan instead, if you have chronic kidney disease.

If the scans show that the tumor has gotten smaller, you will meet with the surgeon to discuss surgery to remove the tumor. If you are scheduled to have surgery, you will stop taking nilotinib 1 day before your surgery date. If the tumor has gotten bigger, you will be taken off study treatment, and other treatment options will be discussed with you. If the scan shows that the tumor is unchanged, you will continue to receive nilotinib until the tumor either shrinks (and you are able to have surgery) or gets bigger (and you are taken off study treatment).

Tumor tissue that is removed during your scheduled biopsy or during surgery will also be used for biological and genetic testing.

After you have surgery, you will receive standard of care treatment off-study, depending on the results of the surgery.

Your doctor may recommend that you begin taking imatinib mesylate after surgery (or if the disease has gotten worse and you are not able to have surgery). In many cases, imatinib mesylate is given on a daily basis for 1-2 years to lower the risk of the disease coming back. During the time after the surgery, information will be collected about your overall health.

If the disease gets worse while you are on study, and you agree, you will be asked to have a tumor biopsy of an easily accessible area. If this happens, this procedure will be described to you in more detail, and you will sign a separate consent.

An assigned research nurse will see you at each clinic visit and will serve as the first contact for any questions or concerns. During the course of this study, you will be asked to report any serious problems or concerns at each study visit. If you have concerns or questions between each study visits, you may contact your study nurse through the Sarcoma Center at M.D. Anderson.

Arm 2 Study Visits:

Participants in Arm 2 will have the following tests and procedures performed:

On Day -7, you will begin taking nilotinib.

On Day -1:

* You will have a a dynamic CT scan within 36 hours before your biopsy to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 0:

-You will have a tumor tissue biopsy performed. To collect a tumor tissue biopsy, the skin above and around the tumor area is numbed with anesthetic, and a sample of tumor tissue is withdrawn through a large needle.

On Day 56:

* You will be asked about your health, any drugs you may be taking, and any side effects you may have experienced.
* You will have a physical exam, including measurement of vital signs and weight.
* Your performance status will be recorded.
* You will have a chest x-ray.
* You will have a standard CT scan or an MRI scan to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

Depending on the results of the tests at Day 56 you will either have surgery, continue nilotinib, or be taken off study and switched to another therapy.

Every 3 months:

* You will be asked about your health, any drugs you may be taking, and any side effects you may have experienced.
* You will have a physical exam, including measurement of vital signs and weight.
* Your performance status will be measured.
* You will have a standard CT scan or an MRI scan to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests.

Additional Testing for Both Groups:

You will have blood (about 1 teaspoon each time) drawn for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. These PK samples will be drawn after the first 6 days of nilotinib (Day -1) and either at the end-of-treatment visit or at any point that the disease gets worse.

When/if your treatment is interrupted for any reason and/or your dose is changed in any way, you will also have ECGs performed. You will have an additional ECG 7 days after this.

End-of-Treatment Visit:

At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You performance status will be recorded.
* You will be asked about your health, any drugs you may be taking, and any side effects you may have experienced.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have an ECG.
* You will have a CT or MRI scan to check the status of the disease.

Length of Study:

You may continue taking the study drug for 1 week (Arm 1) before you have surgery. You may continue taking the study drug for as long as your doctor thinks it is in your best interest, or until you are able to have surgery (Arm 2). You will no longer be able to take the study drug if the disease gets worse or intolerable side effects occur.

Follow-up Testing:

You will be asked to return to the clinic every 3 months for standard follow-up testing, including routine blood tests and CT scans.

This is an investigational study. Nilotinib is FDA approved and commercially available for the treatment of certain types of chronic myeloid leukemia. Its use in patients with GIST is investigational.

Up to 24 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent form must be completed before beginning any study procedure. In order to meet the proposed scientific endpoints, a tissue biopsy will be required at entry. The patient has the right to refuse participation in this study. The ease and ability of the biopsy will be an essential component of the selection process.
2. Continued from #1- Ease and ability of the biopsy will be determined by the enrolling physician and the physician performing the biopsy. The risks and potential complications of biopsy will be explained to each individual patient, with consideration of tumor location, potential damage to nearby organs, potential effect on the patients' quality of life, and the potential effect on the patients performance status.
3. Patients must be greater than or equal to 18 years of age.
4. Histologically documented diagnosis of primary, recurrent, locally advanced and/or metastatic GIST for which complete surgical resection (R0 or R1) is planned by a MDACC sarcoma surgeon.
5. Immunohistochemical documentation of c-kit expression by the tumor.
6. At least one measurable site of disease greater than 1 cm that can be accurately measured in one dimension by plain radiograph, CT, or MRI.
7. Performance status 0, 1, or 2 (ECOG)
8. Adequate end organ function, defined as the following: total bilirubin < 1.5 x ULN (Does not apply to patients with isolated hyperbilirubinemia (e.g. Gilbert's disease) grade <3), ALT and AST < 2.5 x ULN, creatinine < 1.5 x ULN, ANC > 1.5 x 10^9/L, platelets > 100 x 10^9/L, Serum amylase and lipase </ = 1.5 x ULN, Alkaline Phosphatase </= 2.5 x ULN
9. Patients must have the following laboratory values (WNL = within normal limits at the local institution lab) or corrected to within normal limits with supplements prior to the first dose of study medication: Potassium, Magnesium, Phosphorus, Calcium
10. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Female patients who have been surgically sterilized(ie., tubal ligation) should be considered non- childbearing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
11. Written, voluntary informed consent.

Exclusion Criteria:

1. Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
2. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other clinically significant malignant disease which requires systemic treatment (chemotherapy or radiation) is not allowed.
3. Female patients who are pregnant or breast-feeding.
4. Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
5. Patient has a rare hereditary problem of galactose intolerance, severe lactase deficiency or of glucose-galactose malabsorption.
6. Patient with electrolyte abnormality (e.g., hypokalemia, hypomagnesemia, hypophosphatemia, hyperkalemia, hypocalcemia, hyponatremia) unless the level can be corrected to normal levels prior to initiating study drug.
7. Patient has a known brain metastasis
8. Patients with metastasis outside of the peritoneal cavity
9. If patients have any signs or symptoms of metastasis, the appropriate workup should occur prior to enrollment (e.g., CT of the head for a patient with CNS symptoms).
10. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis), acute liver disease, acute or chronic pancreatic disease.
11. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
12. Patient received chemotherapy within 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to study entry, unless the disease is rapidly progressing.
13. Patient with prior exposure to sunitinib, nilotinib or imatinib.
14. Patient previously received radiotherapy to greater than or equal to 25 % of the bone marrow.
15. Patient had a major surgery within 2 weeks prior to study entry.
16. Impaired cardiac function, including any one of the following: Inability to monitor the QT/QTc interval on ECG, Long QT syndrome or a known family history of long QT syndrome, Clinically significant resting bradycardia (<50 beats per minute), QTc > 450 msec on baseline ECG (using the QTcF formula). If QTcF >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc, Myocardial infarction within 12 months prior to starting study
17. Continued from question #16 - Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension defined as greater than 160/100 mmHg despite use of antihypertensive medication), History of or presence of clinically significant ventricular or atrial tachyarrhythmias, Complete left bundle branch block or bifascicular block (right bundle branch block plus left anterior hemiblock) or use of ventricular-paced pacemaker
18. Patients who are currently receiving treatment with any of the medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug
19. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01

PRIMARY OUTCOMES:
Percent of Apoptotic Tumor Cells Pre- and 7 Days Post Nilotinib Treatment | Pre treatment assessment to 7 days post treatment.
  Changes assessed by tumor cell apoptosis measured by Terminal deoxynucleotidyl transferase dUTP nick end labeling (TUNEL) assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Trent, MD, PHD, BS, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org